CLINICAL TRIAL: NCT06301529
Title: The Efficacy and Tolerability of Canagliflozin in Healthy Individuals Comparing Dosing Protocols of Canagliflozin for Use as a Gerotherapeutic
Brief Title: The Efficacy and Tolerability of Canagliflozin in Healthy Individual
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AgelessRx (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ALRx008
Record Dates: First submitted 2024-03-04; First posted 2024-03-08 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Healthy Aging
MeSH Terms: interventions — Canagliflozin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 100mg (Active Comparator): Participants assigned to this arm will be taking 100mg daily, up to 7 times, for study duration.
  Interventions: Drug: Invokana Pill
- 150mg (Experimental): Participants assigned to this arm will be taking 150mg, every other day, up to 4 times, for study duration.
  Interventions: Drug: Invokana Pill

INTERVENTIONS:
Drug: Invokana Pill — 100 mg and 150 mg doses, taken every day and every-other day, respectively.
  Other Names: Canagliflozin

SUMMARY:
The primary objective is to measure the effects that canagliflozin intervention has on reducing average glucose in healthy individuals.

The secondary objective is to assess the tolerability and side effects and urinary glucose excretion following the pulsatile dosing protocol.

DETAILED DESCRIPTION:
This study is designed to mitigate the effects of glucose with intermittent oral Canagliflozin for healthy, non-diabetic volunteers of any sex who enroll in the study. Participants will provide informed consent via AgelessRx electronic medical record. If eligible, prescriptions will be provided online through the AgelessRx website (www.agelessrx.com). Participants will be randomized into two arms: Arm A will take 100 mg of canagliflozin each day for a total of 7 doses, while Arm B will take 150 mg of canagliflozin every other day for a total of 4 doses. Participants in Arm B will also be provided a pill cutter to use throughout the trial on the 300mg tablet.

All participants will begin the trial on the day that they apply a continuous glucose monitor (considered Day 0) and will be asked to take daily blood pressure reading. After one week of baseline readings, both arms will start their canagliflozin dosing protocols.

Participants will be asked to complete 7 total surveys to outline side effects and tolerability, one each day starting after their canagliflozin consumption.

Participants will be asked to complete a dietary intake journal through Day 0 -Day 14. Lifesum (https://lifesum.com/) should be used to track Carbohydrate/Protein/Fat consumption. Participants will share their dietary intake journal twice over their participation (Day 7 & Day 14).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-85
2. Any sex
3. Any ethnicity
4. Interest in taking Canagliflozin
5. Approved by the AgelessRx Medical team to take Canagliflozin
6. Willing and technically able to use and operate a continuous glucose monitor
7. Own a CGM-compatible phone
8. Relatively good health with only well-managed chronic diseases (hypertension, coronary artery disease, type II diabetes, etc.) clinically stable
9. Adequate cognitive function to be able to give informed consent

Exclusion Criteria:

1. Diabetes of any type
2. Taking metformin or any other glucose-lowering medication
3. Other diabetes medication
4. Active malignancy of any kind
5. Clinically relevant renal or kidney disease or dysfunction
6. History of eating disorder
7. Any diuretic
8. Taking any medication, or having any medical condition, that might interfere with the action of canagliflozin or the CGM sensor

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-02-12 (Actual); Primary Completion 2024-06-29 (Actual); Study Completion 2024-06-29 (Actual)

PRIMARY OUTCOMES:
Change in blood glucose values after taking Canagliflozin | 2- weeks
  The primary endpoint, average glucose, will be assessed by examining blood glucose (mg/dL) area under curve as measured by CGM. Glucose data on days without Canagliflozin treatment will serve as a control.

SECONDARY OUTCOMES:
Number of participants with treatment-related side effects through collected survey responses | 2-weeks
  The secondary endpoints of safety and tolerability and urinary glucose excretion will also be assessed. Safety and tolerability will be measured by adverse event reporting, blood pressure monitoring, and by comparing treatment tolerability survey results with control tolerability results through subjective surveys. Urinary glucose excretion will be measured by at-home glucose testing strips.

CONTACTS AND LOCATIONS:
Overall Officials: James P Faber, Study Chair — Institutional Review Board (IRB) of the Institute of Regenerative and Cellular Medicine (IRCM); Sajad Zalzala, MD, Principal Investigator — AgelessRx
Locations (1):
- AgelessRx, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lin HJ, Lee BC, Ho YL, Lin YH, Chen CY, Hsu HC, Lin MS, Chien KL, Chen MF. Postprandial glucose improves the risk prediction of cardiovascular death beyond the metabolic syndrome in the nondiabetic population. Diabetes Care. 2009 Sep;32(9):1721-6. doi: 10.2337/dc08-2337. Epub 2009 Jun 5. PMID 19502543
- [Background] Leiter LA, Yoon KH, Arias P, Langslet G, Xie J, Balis DA, Millington D, Vercruysse F, Canovatchel W, Meininger G. Canagliflozin provides durable glycemic improvements and body weight reduction over 104 weeks versus glimepiride in patients with type 2 diabetes on metformin: a randomized, double-blind, phase 3 study. Diabetes Care. 2015 Mar;38(3):355-64. doi: 10.2337/dc13-2762. Epub 2014 Sep 9. PMID 25205142
- [Background] Suh S, Kim JH. Glycemic Variability: How Do We Measure It and Why Is It Important? Diabetes Metab J. 2015 Aug;39(4):273-82. doi: 10.4093/dmj.2015.39.4.273. PMID 26301188
- [Result] Prasanna Kumar KM, Ghosh S, Canovatchel W, Garodia N, Rajashekar S. A review of clinical efficacy and safety of canagliflozin 300 mg in the management of patients with type 2 diabetes mellitus. Indian J Endocrinol Metab. 2017 Jan-Feb;21(1):196-209. doi: 10.4103/2230-8210.196016. PMID 28217522
- [Result] Papanikolaou Y, Palmer H, Binns MA, Jenkins DJ, Greenwood CE. Better cognitive performance following a low-glycaemic-index compared with a high-glycaemic-index carbohydrate meal in adults with type 2 diabetes. Diabetologia. 2006 May;49(5):855-62. doi: 10.1007/s00125-006-0183-x. Epub 2006 Mar 1. PMID 16508776
- See also: Gottfried, Sara MD, "8 Reason Why Glucose is Worth Measuring." Metabolic Basics. June 17, 2022 — https://www.levelshealth.com/blog/8-reasons-glucose-is-worth-measuring
- See also: Hall H, Perelman D, Breschi A, Limcaoco P, Kellogg R, McLaughlin T, et al. (2018) Glucotypes reveal new patterns of glucose dysregulation. PLoS Biol 16(7): e2005143 — https://doi.org/10.1371/journal.pbio.2005143
- See also: (2022), Canagliflozin and Kidney-Related Adverse Events in Type 2 Diabetes and CKD: Findings From the — https://linkinghub.elsevier.com/retrieve/pii/S0272638621006260

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-01-24): https://cdn.clinicaltrials.gov/large-docs/29/NCT06301529/Prot_SAP_ICF_000.pdf